CLINICAL TRIAL: NCT03858036
Title: Comparison of Corneal Collagen Cross-Linking Performed With "Epi-ON" Versus "Epi-OFF" Techniques in Eyes With Keratoconus and Other Corneal Ectatic Disorders
Brief Title: Corneal Collagen Cross-Linking (CXL) Performed With "Epi-ON" Versus "Epi-OFF" in Eyes With Keratoconus and Other Corneal Ectatic Disorders
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Center for Sight, Sacramento, CA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFS-CXL-001
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Keratoconus; Ectasia
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Epi-OFF CXL (Active Comparator): The Epi-ON treatment will be performed without removal of the corneal epithelium. Ricrolin+will be used as the riboflavin formulation for the pre-treatment and irradiation steps of the Epi-ON treatments. The VEGA UV-A light will be used during the irradiation steps of the Epi-ON treatment.
  Interventions: Drug: Ricrolin+; Device: VEGA UV-A system
- Epi-ON CXL (Active Comparator): The Epi-OFF treatment will be performed with removal of the corneal epithelium before the first dose of riboflavin is administered. Ricrolin+ will be used as the riboflavin formulation for the pre-treatment and irradiation steps of the Epi-OFF treatments. The VEGA UV-A light will be used during the irradiation steps of the Epi-OFF treatment.
  Interventions: Drug: Ricrolin+; Device: VEGA UV-A system

INTERVENTIONS:
Drug: Ricrolin+ — 1 to 2 drops of Ricrolin+ will be instilled topically in the eye every 2 minutes for 30 minutes. At the end of the Ricrolin+ pre-treatment period, the eye will be examined at the slit lamp to detect the presence of a yellow flare in the anterior chamber, indicating adequate riboflavin saturation of the corneal tissue. If the yellow flare is not detected, Ricrolin+ will continue to be instilled 1 drop every 2 minutes for an additional 5 to 10 minutes; and the anterior chamber will be rechecked for yellow flare. This process will be repeated as necessary. During the irradiation period, 1 to 2 drops of Ricrolin+ to cover the cornea (in the same manner as during the riboflavin pre-treatment) before the start of irradiation and every 5 minutes during irradiation until irradiation is complete.
Device: VEGA UV-A system — The VEGA light will be administered for 30 minutes. The VEGA light will stop automatically every 5 minutes for Ricrolin+ administration.

SUMMARY:
This is a prospective, randomized, single investigative site study to compare the safety and effectiveness of Epi-OFF CXL treatment (performed using Ricrolin+ and VEGA UV-A system) compared to Epi-ON CXL (performed using Ricrolin+ and VEGA UV-A system) in eyes with keratoconus and other corneal ectatic disorders.Subjects will be randomized to receive the CXL treatment with either the Epi-On or Epi-Off technique.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 12 years of age or older, male or female, of any race.
2. Having a diagnosis of keratoconus or other corneal ectatic disorder.
3. Presence of central or inferior steepening on the topography map.
4. Axial topography consistent with keratoconus or other corneal ectatic disorder.
5. For eyes diagnosed with keratoconus, presence of one or more slit lamp findings associated with keratoconus, such as:

   1. Scissoring of the retinoscopic reflex
   2. Fleischer ring
   3. Vogt striae
   4. Corneal thinning e .Corneal scarring
6. BSCVA 20/20 or worse.
7. Subject is willing to have CXL performed by the Epi-OFF or Epi-ON techniques.
8. Provide written informed consent and a signed HIPPA form. Pediatric subjects less than 14 years of age must sign an assent and a parent or legal guardian must sign an informed consent.
9. Willingness and ability to follow all instructions and comply with schedule for follow-up visits.
10. If female and capable of becoming pregnant, must not be lactating or pregnant and must agree to use a medically acceptable form of birth control for at least one week prior to the treatment visit and to continue o one month following treatment.

Exclusion Criteria:

1. One of the randomized CXL techniques (Epi-OFF or Epi-ON) is contraindicated or, in the investigator's clinical judgment, is not able to be performed in the study eye.
2. Study eye keratoconus severity is classified as being normal or atypical normal based on the OPD-Scan III keratoconus classification indices.
3. A history of previous corneal transplant in the study eye.
4. A history of prior CXL in the study eye.
5. Corneal pachymetry < 375 microns at the thinnest point as measured by ultrasound pachymetry in the study eye before epithelium removal. [NOTE: Eyes with corneal pachymetry between <375 microns and 325 microns may be enrolled in the compassionate use group.]
6. Presence of Intacs or corneal rings or segments in the study eye.
7. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications or prevent the possibility of improved vision, for example:

   1. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, or corneal dystrophy, etc.)
   2. Clinically significant corneal scarring in the treatment zone unrelated to keratoconus.
8. Eyes which are aphakic.
9. Eyes which are pseudophakic and do not have a UV blocking lens implanted.
10. A known contraindication, sensitivity, or allergy to the test article or its components or to study medications.
11. Nystagmus or any other condition that would prevent a steady gaze during the cross-linking treatment or other diagnostic tests.
12. If female, pregnant, nursing or planning a pregnancy, or having a positive urine pregnancy test prior to the randomization of, or treatment of, either eye during the course of the study.
13. A condition that, in the investigator's opinion, would interfere with or prolong epithelial healing, including a history of chemical injury or delayed epithelial healing in the study eye.
14. Presence or history or any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for cross-linking or study participation or may confound the outcome of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2019-03-08 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in corneal curvature | Baseline, 6 Months, and 12 Months
  Percentage of eyes that had a greater than 2D increase in Kmax measured by the OPD-Scan III

SECONDARY OUTCOMES:
Change in manifest refraction spherical equivalent | Baseline, 6 Months, and 12 Months
  Change in refraction
Change in best-corrected visual acuity (BSCVA) | Baseline, 6 Months, and 12 Months
  Percentage of eyes that had a loss of 2 or more lines in BSCVA
Change in uncorrected-visual acuity (UCVA) | Baseline, 6 Months, and 12 Months
Change in thinnest pachymetry | Baseline, 6 Months, and 12 Months
  measured by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sight, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No